CLINICAL TRIAL: NCT07174323
Title: The Effects of Nextida-GC and Whey Protein on Postprandial Glycemic and Insulinemic Responses When Given 30min Before, 10min Before or With a Standardized Breakfast Test-meal in Healthy Adults With and Without Prediabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: INQUIS Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INQ-2504
Record Dates: First submitted 2025-09-12; First posted 2025-09-15 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Prediabetes; Normal Plasma Glucose; Normoglycemia
Keywords: Glucose; Insulin; prediabetes; whey protein; collagen protein; preload
MeSH Terms: conditions — Prediabetic State; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Those measuring glucose and insulin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- -30 min (Active Comparator): 10 g protein 30 min before eating
  Interventions: Dietary Supplement: Peptide derived from collagen protein; Dietary Supplement: Whey protein isolate
- -10 minutes (Active Comparator): 10 g protein 10 min before eating
  Interventions: Dietary Supplement: Peptide derived from collagen protein; Dietary Supplement: Whey protein isolate
- Control (Sham Comparator): •200 ml water with no protein
  Interventions: Dietary Supplement: Peptide derived from collagen protein; Dietary Supplement: Whey protein isolate
- 0 minutes (Active Comparator): 10 g protein with test meal
  Interventions: Dietary Supplement: Peptide derived from collagen protein; Dietary Supplement: Whey protein isolate

INTERVENTIONS:
Dietary Supplement: Peptide derived from collagen protein — Peptide derived from collagen protein
Dietary Supplement: Whey protein isolate — Whey protein isolate

SUMMARY:
The goals of this clinical trial are to learn if Nextida-GC (a peptide derived from collagen) will reduce postprandial glucose responses when taken 30 minutes before, 10 minutes before or with the first bite of a breakfast test-meal consisting or bread, margarine and jam with a drink coffee, tea or water (each subject will choose a drink and have the same drink each time).

The main questions it aims to answer are:

Does Nextida-GC reduce glucose responses more than whey protein?

What are the effects of Nextida-GC and whey protein on plasma glucose and serum insulin responses when given 30 minutes before eating, 10 minutes before eating, or with the breakfast test meal?

Overall, is it better to take Nextida-GC 30 minutes before eating, 10 minutes before eating, or with the breakfast test meal?

Participants will:

Come to the research center (INQUIS Clinical Research, Toronto, Ontario, Canada) on 8 separate occasions (with bewteen 3 and 14 days between visits) after an overnight fast of at least 10 hours. Each participant will undergo all 8 treatments (one treatment per visit):

Block 1

* 10 grams Nextida-GC in water 30 minutes before eating the test-meal
* 10 grams Nextida-GC in water 10 minutes before eating the test-meal
* water 30min before eating and 10g Nextida-GC in water with the test-meal
* water 30min before eating, and water with the test-meal

Block 2

* 10 grams whey protein in water 30 minutes before eating the test-meal
* 10 grams whey protein in water 10 minutes before eating the test-meal
* water 30min before eating and 10g whey protein in water with the test-meal
* water 30min before eating, and water with the test-meal

The order of the blocks will be randomized and the order of the treatments within the blocks will be randomized.

On each occasions finger-stick blood samples for measuring glucose and insulin will be obtained 30, 10 and 0 minutes before starting to eat the test-meal and 15, 30, 45, 60, 90, 120 and 180 minutes after the first bite of the test-meal.

The main outcome of the study is the area under the curve of plasma glucose from 0 to 180 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant, non-lactating.
* BMI 18.5 to 35.0 kg/m² inclusive.
* n=20 with prediabetes: fasting glucose 5.6-6.9 mmol/L and/or HbA1c 5.7-6.4%.
* n=12 without prediabetes: fasting glucose <5.6 mmol/L and HbA1c <5.7%.
* Systolic blood pressure <160mmHg and diastolic blood pressure <100mmHg.
* Willing to abstain from unusual strenuous exercise and consuming alcoholic drinks for 24 hours before study days.
* Willing to refrain from smoking tobacco or using marijuana in any form (including but not limited to smoking, vaping, edibles, tinctures, or other ingestible or inhalable preparations) for 12h before and during study visits.
* Willing to consume study products that contain animal derived ingredients
* Understand the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator.
* Eligible to receive income in Canada and covered by a health insurance plan such as OHIP.

Exclusion Criteria:

* Failure to meet any one of the inclusion criteria.
* Major trauma or surgical event within 3 months of screening.
* Use of supplements containing collagen and/or high dose of chromium (>500mcg).
* The presence of any laboratory result, health condition, illness or drug use that increases risk to the subject or to others or may affect the results, as judged by the Qualified Investigator.
* Unwillingness or inability to comply with experimental procedures and to follow INQUIS safety guidelines.
* Known intolerance, sensitivity, or allergy to any ingredients in the study test meals.
* Subject is currently participating or recently (within 30 days of screening) participated in a clinical trial involving long-term exposure (greater than 24 hours) to an investigational drug, nutritional supplement, or lifestyle modification

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2026-01-28 (Estimated); Study Completion 2026-01-28 (Estimated)

PRIMARY OUTCOMES:
Glucose iAUC 0-180 | 0 min to 180 minutes
  Incremental area under the glucose curve (iAUC), ignoring area below the concentration at 0 min (just before starting to eat), calculated from plasma glucose measured at 15, 30, 45, 60, 90, 120 and 180 min after starting to eat.

SECONDARY OUTCOMES:
Insulin AUC 0-180 | 0-180 minutes
  Incremental area under the insulin curve (iAUC), ignoring area below the concentration at 0 min (just before starting to eat), calculated from serum insulin measured at 15, 30, 45, 60, 90, 120 and 180 min after starting to eat.
Glucose Peak Rise | 0-180 minutes
  Maximum glucose concentration minus glucose concentration at 0 minutes.
Insulin Peak Rise | 0-180 minutes
  Maximum insulin concentration minus concentration at 0 min.
MAGE | 0-180 minutes
  Maximum Amplitude of Glycemic Excursion measured as the difference between the highest and lowest plasma glucose concentrations.
Glucose Time In Range (TIR) | 0-180 min
  The percent of time when plasma glucose is between 10.0 and 3.9 mmol/L, inclusive (plasma glucose measured at 0, 15, 30, 45, 60, 90, 120 and 180 minutes).
Glucose Time Over Range (TOR) | 0-180 min
  The percent of time when plasma glucose is over 10.0 mmol/L, (plasma glucose measured at 0, 15, 30, 45, 60, 90, 120 and 180 minutes).
Glucose Time Below Range (TBR) | 0-180 min
  The percent of time when plasma glucose is below 3.9 mmol/L, inclusive (plasma glucose measured at 0, 15, 30, 45, 60, 90, 120 and 180 minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wolever, PhD, DM, Principal Investigator — INQUIS Clinical Research
Locations (1):
- INQUIS Clinical Research, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided